CLINICAL TRIAL: NCT06041698
Title: Testing Two Implementation Strategies in Collecting ePRO Among Multiple Myeloma Patients: ePRO4MM
Brief Title: Two Implementation Strategies for the Collection of Electronic Patient-Reported Outcomes Among Patients With Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: iRISID-2022-1329; JT 29004 (Other: JeffTrial Number)
Record Dates: First submitted 2023-08-18; First posted 2023-09-18 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Behavior Therapy; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (TXT-Chatbot ) (Experimental): Patients receive a text message notification and complete surveys through TXT-Chatbot Q2W for 6 months.
  Interventions: Other: Planned Notification; Other: Survey Administration; Behavioral: Behavioral Intervention; Other: Electronic Health Record Review; Other: Interview
- Group II (MyChart/Patient Portal) (Experimental): Patients receive an email notification and complete surveys through MyChart/Patient Portal Q2W for 6 weeks.
  Interventions: Other: Survey Administration; Other: Planned Notification; Behavioral: Behavioral Intervention; Other: Electronic Health Record Review; Other: Interview

INTERVENTIONS:
Other: Planned Notification — Receive text notification
  Other Names: PlannedNotification
  Arms: Group I (TXT-Chatbot )
Other: Survey Administration — Complete surveys
  Arms: Group I (TXT-Chatbot )
Behavioral: Behavioral Intervention — Participate in TXT-Chatbot
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Group I (TXT-Chatbot )
Other: Electronic Health Record Review — Ancillary studies
  Arms: Group I (TXT-Chatbot )
Other: Interview — Ancillary studies
  Arms: Group I (TXT-Chatbot )
Other: Survey Administration — Complete surveys
  Arms: Group II (MyChart/Patient Portal)
Other: Planned Notification — Receive email notification
  Other Names: PlannedNotification
  Arms: Group II (MyChart/Patient Portal)
Behavioral: Behavioral Intervention — Participate in MyChart/Patient Portal
  Other Names: Behavior Conditioning Therapy; behavior modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; BEHAVIORAL THERAPY; Behavioral Treatment; Behavioral Treatments
  Arms: Group II (MyChart/Patient Portal)
Other: Electronic Health Record Review — Ancillary studies
  Arms: Group II (MyChart/Patient Portal)
Other: Interview — Ancillary studies
  Arms: Group II (MyChart/Patient Portal)

SUMMARY:
This clinical trial evaluates satisfaction and engagement with a text messaging platform (TXT-Chatbot) compared to a patient portal system (MyChart/Patient Portal) for reporting symptoms among patients with multiple myeloma (MM). Multiple myeloma is the third most common hematologic (relating to the blood and blood-forming organs) cancer. Patients with MM typically receive continuous therapy from the time of diagnosis, which often comes with treatment-related toxicities. Symptom burden and health-related quality of life (HRQOL) for those with MM can be quite poor. Effects of MM and its treatment may impact HRQOL domains such as physical and emotional well-being, social functioning, and financial burden. Assessment of toxicities through patient-reported outcome (PRO) measures is critical and can generate information to help facilitate clinical decision making and follow up care. PROs are direct reports from patients about their health status. Compared with paper versions, electronic PROs (ePRO) allow patients to report their symptoms in real time outside of their clinic visit, facilitate direct data collection through the electronic health record, and enable clinicians to track symptoms long-term. The use of ePROs is associated with improved patient health outcomes, including better quality of life, reduced emergency department usage, and prolonged overall survival. The increased use of electronic communication technologies to capture PRO data long-term has been implemented through various methods including web-based, social media, text messages, mobile applications, and electronic portals. Text messaging is an accessible, though under-explored, communication channel for promoting ePRO collection. Information gathered from this study may help researchers understand MM patients' preferences for reporting symptoms via text message compared to a patient portal system.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the patients' preference of TXT-Chatbot approach versus MyChart/Patient Portal approach, considering their demographic information.

II. To evaluate each patient's adherence to the approach of his/her own choice by examining their utilization of the ePRO.

SECONDARY OBJECTIVE:

I. To examine the usability and satisfaction of the two implementation approaches of each patient's choice.

EXPLORATORY OBJECTIVE:

I. To explore and measure any differences in patients' preference of TXT-Chatbot approach versus MyChart/Patient Portal approach, as well as the number of completed of ePRO responses, in the course of 6 months, reported between race (African American versus [vs.] Caucasian) and approaches (Chatbot vs. MyChart/Patient Portal).

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP I: Patients receive a text message notification and complete surveys through TXT-Chatbot once every two weeks (Q2W) for 6 months.

GROUP II: Patients receive an email notification and complete surveys through MyChart/Patient Portal Q2W for 6 months.

After completion of study intervention, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MM
* Able to use TXT or have Internet access
* Can read and understand English
* If patients are undergoing an autologous stem cell transplant, they will be enrolled after their transplant

Exclusion Criteria:

* < 18 years of age
* Cognitive impairment documented in the electronic medical record (EMR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the number of completed ePRO responses, assessed in the course of 6 months, based on group. This is a numeric endpoint. | At 6 months
  This is a numeric endpoint.
  For the primary analysis, the number of completed ePRO responses, over the course of 6 months, will be summarized using means and standard deviations, for the two implementation approaches. Multivariable Poisson regression analysis will be performed to explore the relationship between this endpoint and implementation approaches, age, gender, etc., with special consideration of the interaction between race (African American vs. Caucasian) and implementation approaches.

SECONDARY OUTCOMES:
The second endpoint is patients' satisfaction from survey at the end of the intervention. | At 6 months
  The survey contains six (6) questions with Likert scale of responses (very dissatisfied, dissatisfied, neutral, satisfied, very satisfied). A score of 1-5 is assigned to the Likert scales. The overall satisfaction score is defined as the average of scores of the six questions. This is considered as a numeric endpoint.
  For the secondary analysis, the overall satisfaction score with be summarized using means and standard deviations for the two choices of approaches. The dichotomized satisfaction score (overall score >= 3.5) will be summarized using percentages for the two approaches. Multivariable (non-)linear and logistic regression models will be performed to explore the relationship between the endpoints and implementation approaches, age, gender, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States